CLINICAL TRIAL: NCT02274194
Title: Nasal and Oronasal Mask During CPAP Titration on CPAP Level, Apnoea-hypopnoea Index, Airway Defense Biomarkers and Systemic Expression of mi RNA in Patients With Severe Obstructive Sleep Apnea and no History of Nasal Obstruction
Brief Title: Nasal and Oronasal Mask in Severe OSA Patients With Nasal Free Airflow of Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, Associate Professor of Physiotherapy, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 102/13
Record Dates: First submitted 2014-09-30; First posted 2014-10-24 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea of Newborn
Keywords: obstructive sleep apnoea; nasal mask; oronasal mask; breathing route; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal CPAP during titration (Active Comparator): Group nasal mask: use of CPAP for one night whit wash out of two weeks
  Interventions: Device: Nasal CPAP
- Oronasal CPAP during titration (Experimental): Group oronasal mask: use of CPAP for one night with wash out of two weeks.
  Interventions: Device: Oronasal CPAP

INTERVENTIONS:
Device: Nasal CPAP — use of nasal mask to titrate CPAP during a manual full night: if nasal mask is the best interface during titration compared with oronasal mask - patients will go 30-day period of treatment
  Other Names: Nasal mask
  Arms: Nasal CPAP during titration
Device: Oronasal CPAP — use of oronasal mask to titrate CPAP during a manual full night: if oronasal mask is the best interface during titration compared with nasal mask - patients will go 30-day period of treatment
  Other Names: Oronasal mask
  Arms: Oronasal CPAP during titration

SUMMARY:
The obstructive sleep apnea (OSA) affects between 10% to 25% of the adults. Continuous positive airway pressure (CPAP) is the first choice of treatment in severe OSA. However, the adherence to CPAP varies, and the interface between patient and the CPAP may interfere with adherence, comfort and efficiency as well as in sleep variables. Objectives: (1) to determine if self-reported airflow route (nasal or oronasal airflow) is the same as the route determined in a laboratory analysis in controls (healthy subjects) and severe OSA patients with nasal free airflow of obstruction during asleep and awake, (2) to compare the effects of nasal and oronasal CPAP titration (randomized order of masks, 14 days apart) on apnoea-hypopnoea index, CPAP level, PSG variables - including analysis for body positioning, the airway defense mechanisms (nasal mucociliary clearance, mucus properties, citology and inflammation in nasal lavage fluid) and systemic effects (serum miRNA expression and cytokines), (3) CPAP adherence after 1 month and 12 months.

DETAILED DESCRIPTION:
After agreement with the written informed consent, 30 volunteers (10 healthy volunteers and 20 patients with severe OSA), male and female, aged > 21 years were recruited in the Sleep Laboratory of Hospital das Clínicas da Faculdade de Medicina (FMUSP). The volunteers were evaluated at the Sleep Laboratory (Incor) in two phases. First Phase: volunteers were assessed for breathing route awake and asleep (including respiratory events in OSA patients) and were indicated as nasal breathing and oronasal breathing. Second phase for OSA patients: two manual full-night CPAP titration with nasal and oronasal masks in a randomized order, 14 days apart. Data and fluids were analyzed before and after both titration studies comparing both masks including supine and lateral position during asleep and CPAP titration. Third phase for OSA patiens: patients were treated with the best interface found in CPAP titration study during 30 days and patients were assessed for sleep quality, excessive sonolence during the day, airway symptoms, airway defense mechanisms biomarkers (mucociliary clearance, mucus properties, citology, inflammation cytokines and adhesion molecules and others) and serum cytokines and miRNA.

ELIGIBILITY:
Inclusion Criteria:

* >21 years
* moderate or severe obstructive sleep apnea
* nonsmokers
* ex smokers (cessation >12 months)

Exclusion Criteria:

* infection / acute respiratory inflammation (30 days after to study entry)
* history of fixed nasal obstruction
* nasal or upper airways surgery
* chronic diseases without optimized treatment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in Apnea-Hypopnea Index | Baseline (Time 0), after CPAP titration with nasal and oronasal mask (one night with wash out of two weeks) and after 30-day period of treatment
  A full-night diagnostic polysomnography (PSG) was performed in each subject to determine the stages of sleep, an electroencephalogram, electro-oculogram and electromyogram of the submentalis muscle were obtained. Peripheric blood oxygenation was recorded with the use of a finger pulse oximeter. Thoracoabdominal excursions were measured qualitatively using respiratory effort sensors placed over the ribcage and abdomen. Snoring was detected with a vibration snore sensor and body posture with a body position sensor. Subjects used a molded single-piece translucent silicone rubber mask. During titration, a mask with CPAP was added and the procedure was performed according to AASM guidelines.

SECONDARY OUTCOMES:
Airway inflammation by exhaled breath condensate pH | Participants will be assessed at baseline (Time 0), nasal CPAP, oronasal CPAP and after 30-day CPAP treatment (30 days)
  The EBC sample was collected over 15 min of quiet and normal breathings (regular tidal volumes and respiratory rate) through a mouthpiece that was connected to a collector device. Participants were asked to avoid to eat green vegetables and canned or embebbed food the 24 hours before measurements. Ph measurements were performed after dearation with ultrapure argon gas (99.9%).
Nasal mucociliary clearance by saccharine transit time | Participants were assessed at at baseline (Time 0), nasal CPAP, oronasal CPAP and after 30-day CPAP treatment (30 days)
  We evaluate the nasal MCC by measuring nasal saccharine transport time (STT). The subject was asked to avoid alcohol, tea and coffee for 6 hours and to eat or drink nothing for 2 hours before the measurements. The STT assessment is performed in a quiet room at a temperature of 21-22ºC and relative humidity of 63-71%. Subjects sat in a chair and are asked to maintain regular breathing, to avoid deep breathing, coughing, sneezing, sniffing or talking during STT measurements. Twenty-five µg saccharin particles are deposited 2 cm from the anterior end of the non-obstructed nostril and the timer is stopped at the first perception of sweet taste. The maximum delay between the deposition and perception is set at 60 minutes for non-detection.
Nasal inflammation by pH, citology and cytokines and adhesion molecules in nasal lavage | Participants were assessed at baseline (Time 0) and after nasal titration, oronasal titration and CPAP treatment (30 days)
  TNF-α, IL-1beta, IL-6, IL-8, IL-10, IL-13, IL-17, MPO, MIPs, MMPs and cardiovascular panels (multiplex bead assay, Millipore, USA) using ELISA in nasal lavage.
Sleep quality by Pittsburg Questionnaire | Participants will be assessed at at baseline (Time 0) and after CPAP treatment (30 days)
  It is a questionnaire to assess the quality of sleep (basically 7 components) - cut off >5: the worst quality
Upper airways symptoms by SNOT20 questionnaire | Participants will be assessed at at baseline (Time 0) and CPAP treatment (30 days)
  This is a questionnaire that aims to assess quality of life of patients with chronic upper airways symptoms
Excessive sonolence during daytime by Epworth Sleepiness Scale | Participants will be assessed at at baseline (Time 0) and CPAP treatment (30 days)
  This is a questionnaire about daytime sleepiness with 8 questions. Cut-off >10: yes

OTHER OUTCOMES:
Cytokines, adhesion molecules and miRNAs in serum | Participants will be assessed at at baseline (Time 0) and CPAP treatment (30 days)
  TNF-α, IL-1beta, IL-6, IL-8, IL-10, IL-13, IL-17, MPO, MIPs, MMPs and cardiovascular panels (multiplex bead assay, Millipore, USA) using ELISA in nasal lavage. For miRNA PCR analysis, RNA was extracted from the blood sample, quantified and analysed.
adherence to CPAP | 1 and 12 months
  we assessed the time use by CPAP device card
CPAP level | CPAP titration with nasal and oronasal mask (one full night for each mask )
  Using two full-nights polysomnography for CPAP titration. To determine the appropriate CPAP level with nasal and oronasal masks
PSG variables | At baseline and after CPAP titration with nasal and oronasal mask (one full night for each)
  All variables were provided by the study with PSG according to AASM guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Juliana A Nascimento, PhD, Principal Investigator — Faculdade de Medicina da Universidade de Sao Paulo; Naomi K Nakagawa, PhD, Study Director — Faculdade de Medicina da Universidade de Sao Paulo; Geraldo Lorenzi-Filho, PhD, Study Chair — Heart Institute - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo
Locations (2):
- Brazil (2):
  - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No